CLINICAL TRIAL: NCT00154258
Title: An Open Extension Study to Phase IIb Study of Clozapine in Patients With Treatment-resistant Schizophrenia
Brief Title: A Long Term Study of Clozapine in Patients With Treatment-resistant Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEX123J1202
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, treatment-resistant, clozapine
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Clozapine
  Other Names: Clozaril

SUMMARY:
Clozapine is an antipsychotic. This open study will evaluate the safety and efficacy of long term treatment of clozapine in patients with treatment-resistant schizophrenia.

DETAILED DESCRIPTION:
Clozapine is an antipsychotic. This open study will evaluate the safety and efficacy of long term treatment of clozapine in patients with treatment-resistant schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Attended the previous Phase IIb (core) study
* Improved during the core study
* No safety issues during the core study

Exclusion Criteria:

* Discontinued the core study
* Pregnant or nursing (lactating) women

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2001-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Adverse events during the long term treatment (until NDA approval) | Baseline to 52 weeks
Vital signs at every 4 weeks | Baseline to 52 weeks
Laboratory tests (hematology: at every 1 - 2 weeks, others: at every 4 weeks) | Baseline to 52 weeks
ECG at every 12 weeks | Baseline to 52 weeks
Echo cardiogram at every 24 weeks | Baseline to 52 weeks

SECONDARY OUTCOMES:
Changes in the symptoms of psychosis at every 8 weeks up to 52 weeks of treatment, thereafter at every 16 weeks | Baseline to 52 weeks
Motor side effects at every 8 weeks up to 52 weeks of treatment, thereafter at every 16 weeks | Baseline to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals